CLINICAL TRIAL: NCT06478667
Title: The Role of Levosimendan as Inotropic Agent in Acute Aluminum Phosphide-induced Cardiotoxicity: A Randomized Controlled Trial
Brief Title: The Role of Levosimendan as Inotropic Agent in Acute Aluminum Phosphide-induced Cardiotoxicity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Levosimendan in AlP
Record Dates: First submitted 2024-06-23; First posted 2024-06-27 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2024-06

CONDITIONS: Acute Myocarditis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Placebo Comparator): will receive the traditional supportive treatment according to (PCC-ASUH) protocol
  • Interventions: Inotropic agent: Dobutamine Vasopressor: norepinephrine N-acetylcysteine: antioxidant Magnesium Sulphate: antiarrhythmic Sodium Bicarbonate Powder and ondansetron hydrocortisone 100 mg every 4-6h
  Interventions: Drug: levosemindan
- levosemindan group (Active Comparator): will receive the traditional supportive treatment without dobutamine as inotropic agent instead levosimendan will be started in bolus dose of 6-12 µg/kg over 10 minutes followed by infusion of 0.05 - 0.2µg/kg/min with adjusting infusion rate according to response and adverse events.
  Interventions: Drug: levosemindan

INTERVENTIONS:
Drug: levosemindan — inotropic agent

SUMMARY:
To evaluate the potential role of levosimendan as an inotropic agent in aluminum phosphide-induced cardiotoxicity

DETAILED DESCRIPTION:
Aluminum phosphide (ALP) is a well-known fumigant known also as rice pill or wheat pill. It is considered an ideal pesticide since it is effective to preserve stored grains against insects and rodents without leaving residues, in addition to its availability and low cost. In Egypt, it has become a common method of suicide over the last few years because it is cheap and easily accessible. Cardiomyocytes are one of the main targets for ALP. ALP-induced cardiotoxicity involves detrimental effects such as direct myocardial tissue damage, hypoperfusion, myocarditis, pericarditis, and arrhythmias leading to circulatory failure. Levosimendan, an inotropic agent, enhances cardiac contractility through calcium sensitization with minimal oxygen demand and, in turn, decreases the risk of arrhythmia. However, limited studies have investigated the role of levosimendan in the treatment of ALP induced cardiotoxicity.

ELIGIBILITY:
Inclusion Criteria:

Patients with acute ALP intoxication admitted to ICU of PCC-ASUH and developed cardiotoxicity with Poisoning Severity Score (PSS) 2 (moderate) or 3 (severe) that led to cardiogenic shock and necessitated administration of vasoactive medications

Exclusion Criteria:

* Pregnant patients
* The presence of pre-existing diseases such as hematologic, pulmonary, hepatic, renal, immunologic, central nervous system, or endocrine system disorders that made patients unsuitable for the present study.
* Patients with underlying cardiac disease and ECG changes, especially prolonged QTc intervals.
* Patients co-ingested drugs or toxins with cardiovascular toxicity.
* Patients had been previously administered with inotropic agent other than agents under the current study as a preconsultation treatment.
* Patients had received any other investigational medicinal products within 30 days or were enrolled in any other interventional trials with the potential to interact with Levosimendan or affect ALP induced cardiotoxicity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
systolic blood pressure | acute phase of myocarditis in 24 hours
  Maintain systolic blood pressure with adequate organ perfusion

CONTACTS AND LOCATIONS:
Locations (1):
- Poison Control Center, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No